CLINICAL TRIAL: NCT05198440
Title: Neuromodulation of Motion Illusions (Vection)
Acronym: NEUROVEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, Thierry Bougerol, MD, Professor, University Hospital, Grenoble
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ID/RCB 2019-A03159-48
Record Dates: First submitted 2021-12-07; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Healthy
Keywords: vection; neuromodulation; rTMS; tACS
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuromodulation of vection (Experimental)
  Interventions: Device: non-invasive neuromodulation; Device: electroencephalography; Device: anatomical MRI

INTERVENTIONS:
Device: non-invasive neuromodulation — The modulations of the vection phenomenon will then be studied over two sessions of 1h30, separated by a minimum of 3 to a maximum of 15 days (the first session will be performed following the MRI). Each session will include: the installation of an EEG headset and the parameterization of the stimulation (30 min), then a phase of recording of the vection with neuromodulation (1h) according to 2 experimental conditions:
  * Experiment 1: recording of vection at rest (20 min), then during and after neurostimulation by tES (20 min). Active and sham (placebo) stimulation will be tested separately during the two sessions (counterbalanced order).
  * Experiment 2: recording of vection during neuromodulation by rTMS triggered in real time (1h). Triggering will be based on behavioral response (experiment 2a) or oscillatory activity detection (experiment 2b). Active and sham (placebo) stimulation will be tested in both sessions (randomized order).
  Other Names: rTMS; tACS
Device: electroencephalography — The modulations of the vection phenomenon will then be studied over two sessions of 1h30, separated by a minimum of 3 to a maximum of 15 days (the first session will be performed following the MRI). Each session will include: the installation of an EEG headset and the parameterization of the stimulation (30 min), then a phase of recording of the vection with neuromodulation (1h) according to 2 experimental conditions:
  * Experiment 1: recording of vection at rest (20 min), then during and after neurostimulation by tES (20 min). Active and sham (placebo) stimulation will be tested separately during the two sessions (counterbalanced order).
  * Experiment 2: recording of vection during neuromodulation by rTMS triggered in real time (1h). Triggering will be based on behavioral response (experiment 2a) or oscillatory activity detection (experiment 2b). Active and sham (placebo) stimulation will be tested in both sessions (randomized order).
  Other Names: EEG
Device: anatomical MRI — The modulations of the vection phenomenon will then be studied over two sessions of 1h30, separated by a minimum of 3 to a maximum of 15 days (the first session will be performed following the MRI). Each session will include: the installation of an EEG headset and the parameterization of the stimulation (30 min), then a phase of recording of the vection with neuromodulation (1h) according to 2 experimental conditions:
  * Experiment 1: recording of vection at rest (20 min), then during and after neurostimulation by tES (20 min). Active and sham (placebo) stimulation will be tested separately during the two sessions (counterbalanced order).
  * Experiment 2: recording of vection during neuromodulation by rTMS triggered in real time (1h). Triggering will be based on behavioral response (experiment 2a) or oscillatory activity detection (experiment 2b). Active and sham (placebo) stimulation will be tested in both sessions (randomized order).

SUMMARY:
Virtual reality systems or simulators are more and more frequently used in the field of learning but also in motor rehabilitation. One of the key points of the success of these systems is the experience of "presence" which is associated with the capacity of these technologies to develop in the observer, who is static, the sensation of moving in the virtual environment (vection). However, the simulation generates a sensory conflict (an optical flow specifying self-motion and vestibular stimuli specifying body immobility). This conflict influences the temporal characteristics of the vection and consequently modifies the way users act in their virtual environment. Thus, contrary to a real situation, vection does not occur instantaneously with the appearance of a visual movement. Moreover, the visual stimulus often generates alternating periods of perception of movement of the environment and of oneself (bistable perception) which can lead to "simulator sickness", a disabling situation for the user. Thus, as vection is an essential element to allow an "optimal transfer of learning" from the simulator to reality, it may be important to promote its emergence while limiting its bistability.

The aim of this project is to study the inhibitory or facilitative modulation of the emergence of the vection phenomenon by the use of non-invasive cortical stimulation techniques (transcranial electrical stimulation (tES), transcranial alternative current stimulation (tACS), and repeated transcranial magnetic stimulation (rTMS)).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 to 40 years
* Right-handed subjects
* Signed informed consent,
* Medical examination performed prior to participation in the research,
* Affiliation to or beneficiary of a social security plan

Exclusion Criteria:

* Contraindications (CI) to the practice of MRI, EEG, TMS & tES
* Existence of a severe general condition: cardiac, respiratory, hematological, renal, hepatic, cancerous,
* Regular use of anxiolytics, sedatives, antidepressants, neuroleptics,
* Characterized psychiatric pathology,
* Ingestion of alcohol before the examination,
* Pregnant, parturient or breastfeeding women
* Person deprived of liberty by judicial or administrative decision, person under a legal protection measure (under guardianship or curators)
* Participation in other interventional research protocols in progress with an exclusion period or in the previous week Subject who would receive more than 4500 euros of compensation due to his participation in other research involving the human person in the 12 months preceding this study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in the latency of first vection between neuromodulations | During the two experimental sessions, at day 1 and up to day 15
  Time required for the appearance of a vection before and after neurostimulation (latency in s).
Change in the vection frequency between neuromodulations | During the two experimental sessions, at day 1 and up to day 15
  Frequency of vection episodes during a period of visual stimulation before and after neurostimulation (%).
Change in the vection duration between neuromodulations | During the two experimental sessions, at day 1 and up to day 15
  Perceived total time experiencing vection during visual stimulation before and after neurostimulation (s).
Change in the vection intensity between neuromodulations | During the two experimental sessions, at day 1 and up to day 15
  Intensity of vection before and after neurostimulation (subjective scale from 0 to 10).

SECONDARY OUTCOMES:
Change in brain activity (as measured by EEG - EP) between neuromodulations | During the two experimental sessions, at day 1 and up to day 15
  - Evoked potentials (V)
Change in brain activity (as measured by EEG - spectrum) between neuromodulations | During the two experimental sessions, at day 1 and up to day 15
  - Oscillatory activity (V^2 / Hz)
Change in brain activity (as measured by EEG - connectivity) between neuromodulations | During the two experimental sessions, at day 1 and up to day 15
  - Functional connectivity (%)